CLINICAL TRIAL: NCT07404800
Title: Longitudinal Investigation of the Risk and Protective Factors of Dating Violence (Dating it Safe) - Firearms
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Rhode Island Hospital (Other); Georgia State University (Other); Sam Houston State University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Temple, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-24-0006; R01CE003614 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dating Violence; Firearm Injury and Violence
Keywords: dating violence; interparental violence; community violence; firearm injury; firearm violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort consists of adult participants with an average age of 28 - 30 years old.

SUMMARY:
This sub-study aims to identify key individual (e.g., demographic, socioeconomic, attitudes), relationship, behavioral and situational, trauma related, and neighborhood/community risk and protective factors for gun access, carriage, and use.

DETAILED DESCRIPTION:
The use of an ongoing longitudinal dataset is cost-effective, efficient, and highly innovative in that we will examine developmental and prospective factors associated with FIV. Indeed, our dataset fills gaps in our existing understanding of FIV through robust assessment of trauma history, risk and protective factors, employment, relationships, and physical and mental health. The study team's use of a community sample, emphasis on protective factors, innovative combination of assessment methods (quantitative and qualitative) and multiple sources (self-reports and official records), and research translation and dissemination to policymakers and practitioners will produce an unparalleled and detailed account of FIV. Findings will be critically important to theoretical development and refinement, as well as informing evidence-based FIV prevention and intervention programs and policy.

ELIGIBILITY:
Inclusion Criteria:

* Waves 1-13 (years 2010-2024): High school freshman and sophomores located at a designated study school and classroom that returned a signed parent consent form and student assent form.
* Beginning with Wave 10, current partners of participants are eligible to participate.
* Waves 13 - 14 (years 2024-2025) + Firearm injury and violence (FIV) cohort: Original study participants from Waves 1-13 and their current partners will be asked gun usage survey questions. Anyone endorsing gun carriage in Wave 11 will be eligible for an in-depth interview in Waves 13 - 14.

Exclusion Criteria:

- Anyone not originally consented in 2010 or not a current partner of a participant originally consented in 2010 is not eligible to participate in the research survey. Participants who declined to participate or passed away during previous waves will not be included. Anyone not endorsing gun carriage in Wave 11 will be excluded from in-depth interview invitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High school freshman and sophomores from 7 ethnically diverse high schools located in Southeast Texas.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Identify key individual (e.g., demographic, socioeconomic, attitudes), relationship, behavioral and situational, trauma related, and neighborhood/community risk and protective factors for gun access, carriage, and use. | From 2024 to 2027
Qualitative interviews with known gun-carriers | 2024-2027
  Conduct a series of 60 in-depth semi-structured interviews with known gun-carriers (Mean age = 26) recruited from Wave 10 of the ongoing study to better understand their thinking, practices, contexts, and experiences of acquiring, carrying, using, sharing, and storing firearms.

OTHER OUTCOMES:
Disseminate evidence based products | 2024-2027
  Taking the complex political environment into account, we will translate results into jargon-free language and disseminate evidence-based products (i.e., policy briefs, summary reports) to policymakers and practitioners to inform FIV prevention legislation.
  By leveraging and extending the scope and breadth of our robust longitudinal dataset and conducting in-depth qualitative interviews of known gun carriers, we will enhance our understanding of the risk and protective factors related to firearm access, carriage, and use. Findings from this mixed-methods project will directly benefit the field by informing policy and the evolution of developmentally appropriate evidence-based interventions, with the ultimate goal of reducing firearm violence among adolescents and young adults.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Temple, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No